CLINICAL TRIAL: NCT02005328
Title: Study of the Effect and Safety of Three New Oral Sprays and a Reference Marketed Oral Spray in the Relief of Drug-induced Xerostomia Associated With Hyposialia.
Brief Title: Exploratory Study in the Relief of Drug-induced Xerostomia Associated With Hyposialia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DC0161 BS 0 01; CIV-13-10-011648 (Other: EUDAMED)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Drug-induced Xerostomia
Keywords: Xerostomia; hyposialia; hyposalivation; saliva substitute; Salivary Gland; Mouth Diseases; Dry mouth
MeSH Terms: conditions — Xerostomia; Mouth Diseases

ARMS (1):
- cross-over (Experimental): Four periods separated by a wash out lasting up to 3 days at maximum. At each period, application of one product (twice). Duration of treatment period: From 4 to 13 days.
  Interventions: Device: Tested product : DC161-DP0291; Device: Tested product : DC161-DP0292; Device: Tested product : DC161-DP0293; Device: Reference product: solution for oromucosal sprays

INTERVENTIONS:
Device: Tested product : DC161-DP0291 — Application of product in the mouth twice daily
Device: Tested product : DC161-DP0292 — Application of product in the mouth twice daily
Device: Tested product : DC161-DP0293 — Application of product in the mouth twice daily
Device: Reference product: solution for oromucosal sprays — Application of product in the mouth twice daily

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy, the safety and acceptability of three new oral sprays with a reference oral spray in the relief of drug-induced xerostomia associated with hyposialia, i.e. dryness of the mouth induced by a decrease of salivation (hyposialia) induced by chronic drug intake.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects,
* Adult subjects (≥18 years) taking drug(s) causing salivary hypofunction / xerostomia, for at least 1 week prior to study initiation and expected to continue without change during study
* Subjects with a complaint of dry mouth as assessed by a response of 40mm or greater on item "Rate the dryness of your mouth" of the Dry Mouth Visual Analogue Scale (VAS) questions. (The VAS limits will be 0 representing normal [i.e. no dry mouth symptoms] and 100 representing "the worst imaginable" dry mouth symptoms). This score should also be met before the 1st product application, on P1 D1.
* Documented hyposalivation with test of resting saliva weight absorbed ≤ 0.5g/5 min at baseline

Exclusion Criteria:

* Presence of disorders (bucco-dental disease, history of major medical/psychiatric illness or surgery, ... ) which, in the judgement of the investigator, may interfere with study implementation and/or study parameter assessment(s).
* Sjögren syndrome and related autoimmune diseases,
* Other medical causes of xerostomia (oral candidiasis).
* History of head and neck irradiation and cancer chemotherapy
* History of hypersensitivity to any of the components of the investigational products,
* History or current excessive use of alcohol,
* History of drug addiction,
* Presence of treatments for their dry mouth within 7 days prior to inclusion into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Observed area under the curve of dry mouth evaluations | 11 points : from baseline (before application) and up to 4 hours after the first product application
  Dry mouth will be self-rated using item "Rate the dryness of your mouth" of the Dry Mouth Visual Analogue Scale questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Erfurt, Germany